CLINICAL TRIAL: NCT04588012
Title: Et Randomiseret Kontrolleret Pilotstudie af OurRelationship.dk, et Online selvhjælpsforløb Til Par Med Mange Konflikter Eller Lav Trivsel i Parforholdet.
Brief Title: A Pilot Study of OurRelationship.dk, a Web-based Self-help-Program for Couples With High Levels of Conflict or Distress
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: TrygFonden, Denmark (Industry); University of Miami (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 72253
Record Dates: First submitted 2020-10-07; First posted 2020-10-19 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-03

CONDITIONS: Relationship Distress; Marital Conflict; Family Relationship

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Online self-help the OurRelationship.dk program (Experimental): Couples in the intervention condition will receive the full OurRelationship program including the three modules, the Observe, the Understand, and the Respond module. The program takes 6-8 hours to complete the program after the randomization. The second coach call will take place after the Observe phase. The third coach call will take place after the Understand phase. The fourth coach call will take place after the Respond phase.
  Interventions: Behavioral: The online self-help Program OurRelationship developed by prof. Brian Doss and prof. Andrew Christensen.
- Off line self-help the book "Pas på Parforholdet" (Active Comparator): Couples in the active control group receive two copies of the book "Pas på parforholdet, når kærligheden er kommet for at blive" [Take care of your relationship when love is here to stay] by Mattias Stølen Due (2016). This book includes general research based knowledge on maintaining a healthy relationship as well as questions and exercises for couples to do on their own. To support couples in an activate self-help approach, a sheet with guidelines on using the book will help couples plan their reading and couple conversations. Regular questionnaires will be sent to couples in the control group (matched timely to the questionnaires received by the intervention group). As such, the active control condition will mirror the benefit that couples are likely to get from using well-chosen, solid literature with the addition of any benefit that the research participation (filling in questionnaire) will generate.
  Interventions: Behavioral: The off line self-help course "Pas på Parforholdet".

INTERVENTIONS:
Behavioral: The online self-help Program OurRelationship developed by prof. Brian Doss and prof. Andrew Christensen. — The OurRelationship program is developed by prof. Brian Doss and prof. Andrew Christensen.
  Arms: Online self-help the OurRelationship.dk program
Behavioral: The off line self-help course "Pas på Parforholdet". — The book "Pas på parforholdet" is written by Mattias Stølen Due.
  Arms: Off line self-help the book "Pas på Parforholdet"

SUMMARY:
The aim of this study is twofold 1) to conduct a pilot test of methods for a larger scale RCT study evaluating the efficacy of OurRelationship offered to couples with high levels of conflict or distress and at least one child at the address, and 2) to test if the OurRelationship program meets predefined feasibility criteria when implemented in a real-world setting. If study results on these two aims are convincing, a full scale RCT of the intervention will be pursued.

DETAILED DESCRIPTION:
A cost-effective online self-help program for distressed couples could help serve more couples, in particular those with limited access to traditional couple therapy. The OurRelationship program, a web-based, primarily self-help program for couples developed in the US, has previously shown medium to large effects sizes on relationship functioning for a diverse sample of couples and these effects were maintained over 12 months (Doss et al., 2016; 2020). These findings promise a large potential in online self-help for couples, if findings replicate in independent research.

For the pilot, 80 couples experiencing high levels of conflict or distress in their relationship and who had at least one child at the address were recruited through a study website (www.ourelationship.dk) build for the pilot. Couples were randomized to receive either the Danish version of the program including 4 coach calls, or an active control condition receiving two copies of a self-help book and a plan for 4 x 30 min couple conversations. In this pilot, research methods in terms of recruitment, randomization, completion of program, test of measures, and data collection are evaluated.

ELIGIBILITY:
Inclusion Criteria:

To detail the criteria "high level of conflict or distress", one or both of the following criteria must be fulfilled:

1. One or both partners report being victim or perpetrator of at least one act of physical or psychological aggression during the past year OR
2. One partner score at least 1 standard deviation (SD) (indicating severe relationship distress) or both partners 0.5 SD below the Danish population mean on a measure for relationship satisfaction (Couple Satisfaction Index; Funk & Rogge, 2007).

In addition:

* both partners in the couple have to be 18 or above
* been living together for at least six months
* have at least one child below 18 years living at home
* be able to read and understand Danish
* have access to the Internet, a tablet, computer, or telephone
* willing to refrain from couple therapy (or other couple interventions) within the period of the project.

Exclusion Criteria:

* Plans on divorcing, breaking up or having an ongoing affair
* Moderate to severe levels of suicidal ideation (>=7 on the Suicidal Behavioral Questionnaire-Revised, Osman et al., 2001)
* Victimization of intimate partner violence resulting in injury or fear within the last three months (using screener items developed by Beach, Whisman, Snyder, & Heyman, 2013).
* Taking psychotropic drugs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — heterosexual couples are eligible for the study
Enrollment: 182 (Actual)
Dates: Start 2020-09-15 (Actual); Primary Completion 2023-02-10 (Actual); Study Completion 2023-02-10 (Actual)

PRIMARY OUTCOMES:
Relationship Satisfaction: Danish 4-item version of the Couple Satisfaction Index | Pre-to-post (time frame spanning across 8 weeks)
  As measured by the Danish 4-item version of the Couple Satisfaction Index (CSI; Funk & Rogge, 2007). A higher score indicate more relationship satisfaction.
Intimacy | Pre-to-post (time frame spanning across 8 weeks)
  "Psychological" intimacy was assessed by four items on 5-point scales. Items were: I felt close to, secure with, cared for, and understood (Debrot et al, 2013). A higher score indicate more intimacy between partners.

SECONDARY OUTCOMES:
Depressive symptoms | Pre-to-post (time frame spanning across 8 weeks)
  As measured by the Major Depression Inventory (Olsen, Jensen, Noerholm, Martiny, & Bech, 2003). A higher score indicate more depressive symptoms.
Relationship Confidence scale | Pre-to-post (time frame spanning across 8 weeks)
  Two items from the Confidence Scale (Rhoades, Stanley, & Markman, 2009). A higher score indicate more confidence.
Positive and Negative Relationship Quality | Pre-to-post (time frame spanning across 8 weeks)
  As measured by the eight-item Positive and Negative Relationship Quality scale (Fincham, & Rogge, 2010). Participants were asked to separately rate four positive (e.g., enjoyable, alive) and four negative (e.g., bad, lifeless) dimensions of their relationship. Higher scores on the positive and lower scores on the negative scale indicate more relationship quality.

CONTACTS AND LOCATIONS:
Overall Officials: Tea L. Trillingsgaard, Ph.D, Principal Investigator — University of Aarhus
Locations (1):
- Aarhus University, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: No